CLINICAL TRIAL: NCT01771003
Title: The Effect of Remote Ischemic Preconditioning in Partial Nephrectomy
Brief Title: Remote Ischemia Pre-Conditioning in Patients Undergoing Partial Nephrectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RIPC
Record Dates: First submitted 2012-10-29; First posted 2013-01-18 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Renal Cell Carcinoma
Keywords: Partial nephrectomy; renal cell carcinoma; Renal Function; Remote ischemia preconditioning
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Without CellAegis' autoRIC™ Device (Placebo Comparator): patients will have a blood pressure cuff attached to their arm that will not inflate/deflate as in the active group
  Interventions: Device: CellAegis' autoRIC™ Device
- With CellAegis' autoRIC™ Device (Active Comparator): Patients will have the CellAegis' autoRIC™ Device attached and it will inflate to 200 mmHg in four 5 minute cycles with intervening 5 minutes of reperfusion with the cuff deflated between cycles (while under general anesthetic)
  Interventions: Device: CellAegis' autoRIC™ Device

INTERVENTIONS:
Device: CellAegis' autoRIC™ Device — Patients in the active group will have the autoRIC device (like a blood pressure cuff) inflated and deflated to a pressure of 200 mmHg in four 5 minute cycles with intervening 5 minutes of reperfusion with the cuff deflated between cycles

SUMMARY:
Partial Nephrectomy has become the standard treatment in patients with tumours <7cm (T1). Even though this is a nephron sparing surgery, there is still potential for acute kidney injury, due to ischemia during the surgery. Remote Ischemia Preconditioning may prevent acute kidney injury and in turn chronic kidney disease. Remote Ischemia pre-conditioning involves applying a blood pressure cuff and inflating and deflating several times immediately prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be a candidate for laparoscopic partial nephrectomy
* ECOG Performance status of 0-1

Exclusion Criteria:

* No diagnosis of any current cutaneous, vascular or neural disease in the right upper arm.
* If the patient received isoflurane for any indication during the operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in Kidney Function before and after surgery | up to 2 weeks prior to surgery and up to 24 hrs post surgery
  To measure and compare kidney function (Cr, eGFR) and AKI biomarkers in patients undergoing partial nephrectomy with and without RIPC

CONTACTS AND LOCATIONS:
Overall Officials: Michael Jewett, M.D., Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada